CLINICAL TRIAL: NCT05096468
Title: Esketamine Combined With Pregabalin on Acute Postoperative Pain in Patients Undergoing Resection of Spinal Neoplasms.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z19110000661906703
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Esketamine; Pregabalin; Acute Postoperative Pain; Neurosurgical Procedures; Perioperative Complication; Spinal Cord Neoplasms
MeSH Terms: conditions — Pain, Postoperative; Spinal Cord Neoplasms | interventions — Esketamine; Pregabalin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine and pregabalin (Experimental)
  Interventions: Drug: S-ketamine and pregabalin
- Normal saline and placebo capsule (Placebo Comparator)
  Interventions: Drug: Normal saline and placebo capsule

INTERVENTIONS:
Drug: S-ketamine and pregabalin — * Drug: Pregabalin
  * 150mg (2hrs) pre operatively and 75mg twice daily post operatively for 7 days(POD1-7), followed by dose reduction to 75mg once daily for 7 days(POD8-14)
  * Drug: S-ketamine infusion
  * 0.5 mg/kg bolus after induction of anesthesia +0.12 mg/kg/h continuous intravenous infusion for 48 h
  Arms: S-ketamine and pregabalin
Drug: Normal saline and placebo capsule — * Drug: Placebo capsules
  * Two placebo capsules (2hrs) preoperatively and twice daily post operatively for 7days, followed by dose reduction to single capsule once daily for 7days
  * Drug: Normal saline
  * 0.9% saline bolus after induction of anesthesia + intravenous infusion for 48 hours
  Arms: Normal saline and placebo capsule

SUMMARY:
Postsurgical pain is now known to be one of the most common and difficult-to-treat complications of surgery. severe postoperative pain can significantly impair patients' quality of life, social functioning and contribute to excessive health care expenditures. It is worth noting that acute postoperative pain may play a vital role in central sensitization and up-regulation of pain receptors, even factors implicated in the development of CPSP. According to previous studies, the incidence of postoperative pain among patients undergoing spinal surgery was nearly 80%. At the same time, perioperative pain management of patients undergoing spinal surgery has not been clearly. For the past few years, pregabalin and esketamine are becoming important roles in perioperative pain management, lots of studies have shown that these two analgesics might relieve postoperative pain. The aim of this study was to evaluate the acute analgesic effects of esketamine and pregabalin in combination after spinal cord neoplasms resection, so as to find a better way to help the patients undergoing spinal surgery keep away from the acute perioperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective spinal cord neoplasms resection;
* Ages between 18 and 65 years old;
* American Society of Anaesthesiology (ASA) status I-III;
* Signed informed consent.

Exclusion Criteria:

* Previous adverse reaction to ketamine, s-ketamine or pregabalin;
* Patients with a diagnosed history of severe chronic pain;
* Patients with long-term analgesic treatment(gabapentin/opioids/ketamine);
* Patients with aphasia or inability to cooperate with the pain assessments;
* Known sever insufficiency of vitals(such as heart failure/renal dysfunction/hepatic failure);
* Patients with a diagnosed history of psychiatric disorder;
* Patients treated with gabapentin/pregabalin in the last three months;
* Drug abuse;
* Body mass index (BMI) > 35 kg/m2 ;
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with acute moderate-to-severe postsurgical pain during 48h after operation | 48 hours after operation
  The primary outcome was the proportion of patients with acute moderate-to-severe postsurgical pain during the 48-h postoperative period (defined as a VAS score ≥ 40 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Derived] Zhou Y, Sun W, Fu Y, Wang J, Fan J, Liang Y, Jia W, Han R. Effect of esketamine combined with pregabalin on acute postsurgical pain in patients who underwent resection of spinal neoplasms: a randomized controlled trial. Pain. 2024 Sep 1;165(9):e96-e105. doi: 10.1097/j.pain.0000000000003211. Epub 2024 Mar 15. PMID 38501980
- [Derived] Sun W, Wang J, Wang J, Fan J, Zhou Y, Wang Y, Han R. Esketamine combined with pregabalin on acute postoperative pain in patients undergoing resection of spinal neoplasms: study protocol for a randomized controlled trial. Trials. 2023 Feb 25;24(1):144. doi: 10.1186/s13063-023-07178-3. PMID 36841794